CLINICAL TRIAL: NCT05099835
Title: Ultrasound-Guided Stellate Ganglion Block With Botulinum Toxin Versus Steroid in Refractory Bell's Palsy
Brief Title: Ultrasound-Guided Stellate Ganglion Block With Botulinum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 000092
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Change From Baseline House-Brackmann
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum Toxin (Active Comparator): injected 10 mL of 0.1% bupivacaine with 100 Botox units (BOTOX®, Allergan Inc., Irvine, CA, USA)
  Interventions: Drug: Botox
- steroid (Active Comparator): injected 10 mL of 0.25% bupivacaine with triamcinolonacetonide 4 mg/ml
  Interventions: Drug: triamcinolonacetonide

INTERVENTIONS:
Drug: Botox — injected 10 mL of 0.1% bupivacaine with 100 Botox units (BOTOX®, Allergan Inc., Irvine, CA, USA)
  Arms: Botulinum Toxin
Drug: triamcinolonacetonide — triamcinolonacetonide stellate ganglion injection
  Arms: steroid

SUMMARY:
the local stellate ganglion block with bupivacaine and corticosteroid treatment for acute peripheral facial nerve palsy in patients can induce hyperglycemia, and an alternative local therapy may be necessary and some time may ve ineffective. Our purpose in this study is to evaluate therapeutic effects of stellate ganglion block (SGB) Botulinum Toxin on referactory facial nerve palsy

DETAILED DESCRIPTION:
:Idiopathic facial nerve palsy (Bell's palsy) is caused by damage to the facial nerve at any site of the peripheral branches after the facial nucleus.Stellate ganglion block is inteneded to increase blood flow and promotes nerve regeneration. the local stellate ganglion block with bupivacaine and corticosteroid treatment for acute peripheral facial nerve palsy in patients can induce hyperglycemia, and an alternative local therapy may be necessary and some time may ve ineffective. Our purpose in this study is to evaluate therapeutic effects of stellate ganglion block (SGB) Botulinum Toxin on referactory facial nerve palsy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by clinical and neurological assessment as one-sided idiopathic facial palsy
* Age 18 to 60 •-ASA i-II

Exclusion Criteria:

* Exclusion Criteria:

  * diabetic
  * coagulation dysfunction
  * mental or cognitive dysfunclion
  * allergy to injected medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline House-Brackmann | : Baseline ,change from baseline House-Brackmann at 7th day,one month,two month, three month
  Change from Baseline House-Brackmann

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No